CLINICAL TRIAL: NCT05911672
Title: Testing and Evaluating the Collection of Patient Reported Outcomes In Cancer CarE Using Innovative Approaches: The ePROM Digital Health Tool
Brief Title: Testing and Evaluating the Collection of Patient Reported Outcomes In Cancer Care Using Innovative Approaches
Acronym: PRICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cyprus University of Technology (Other)
Collaborators: German Oncology Center, Cyprus (Other); CYENS Centre of Excellence (Unknown)
Responsible Party: Principal Investigator, Angelos Kassianos, Lecturer, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CUT_DN_03; OPPORTUNITY/0916/ MSCA/0016 (Other: Cyprus Research and Innovation Foundation)
Record Dates: First submitted 2023-06-08; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Cancer
Keywords: cancer; digital health; Ecologically Momentary Assessment; Ecologically Momentary Intervention; Virtual Reality
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: patients will be randomized into three groups: Full Intervention; Partial Intervention and Control
Who Masked: Participant, Care Provider
Masking Description: Patients and providers (nurses and clinicians) will be blinded on the type of intervention received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full Intervention (Experimental): This group will receive the app (PRICE) which will collect their PROMs (pain, fatigue and stress) three times a day for 2 weeks. They will be prompted each time they have elevated levels of pain, fatigue and stress to use the VR glasses (EMI). This is the EMI provided: https://dl.acm.org/doi/abs/10.1145/3491101.3503562?casa_token=tC5fSN8-k5EAAAAA:56_TMf6HitVQXZypY2j9FCCcroIFZW9kxxzCEt0yJNFJmNrv79m9W7htznSzMWqGLwE4eimBU0vkLA
  Interventions: Device: PRICE
- Partial Intervention (Active Comparator): This group will receive the EMA app and the EMI but they will not be prompted to use the EMI according to their EMA data.
  Interventions: Device: PRICE
- Control (No Intervention): This group will receive the EMA but no the EMI.

INTERVENTIONS:
Device: PRICE — Working closely with 51 cancer patients, medical and paramedical personnel, we co-designed an intelligent personalized mobile application to first collect ecologically momentary assessment data on symptoms like pain and fatigue and Health-Related Quality of Life and subsequently enhance symptom management of cancer patients at home. The full description is available here: https://dl.acm.org/doi/abs/10.1145/3491101.3503562?casa_token=tC5fSN8-k5EAAAAA:56_TMf6HitVQXZypY2j9FCCcroIFZW9kxxzCEt0yJNFJmNrv79m9W7htznSzMWqGLwE4eimBU0vkLA
  Arms: Full Intervention; Partial Intervention

SUMMARY:
Patient Reported Outcome Measures (PROMs) are patients' reports of their symptom experience, quality of life and functionality. These measures are used as an endpoint to clinical trials but rarely integrated into routine cancer care. Moreover, they are resource intensive and prone to retrospective biases. PRICE project aims to develop and evaluate a digital health tool (ePROM), collecting PROMs at the clinic and additional Ecological Momentary Assessment (EMA) of PROMs using a mobile application. In addition it tests whether patients who are identified to have elevated pain, fatigue, and stress will benefit from an Ecological Momentary Intervention (EMI) based on Virtual Reality environments. EMA can overcome biases and barriers in PROM assessment whilst EMI can offer an easy and possibly cost-effective intervention until patients re-visit the clinic. The project can contribute to monitoring patient data and achieve viable health systems. It is also timely since digital health tools are considered the future of oncology care but often lack robustness in development and evaluation. Patients treated for cancer at the German Oncology Centre in Cyprus will be randomized into three conditions: (a) Full Intervention (patients who are prompted to use the EMI based on their EMA data; (b) Partial Intervention (patients who are prompted to use the EMI irrespective of their EMA data); (c) Control (patients who only provide their EMA without an EMI). A dissemination strategy will ensure findings and innovation are available to the public, clinicians, students and policy-makers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with any type of cancer
* Treated as either inpatient or outpatient
* Good understanding of Greek
* Able to consent
* No psychiatric comorbidities

Exclusion Criteria:

* Diagnosed with psychiatric disorders
* Unable to consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in usability and feasibility from baseline to one week later | Baseline, after treatment (1 week later)
  System Usability and Feasibility questionnaire

SECONDARY OUTCOMES:
EORTC QLQ-C-30 | Baseline, after treatment (1 week later)
  Health-Related Quality of Life. Using the global quality of life scale (minimum 0, maximum 100), with higher scores indicating better outcome (higher quality of life)
Fatigue Assessment Scale (FAS) | Baseline, after treatment (1 week later)
  Fatigue Assessment Scale with one score (minimum 10 maximum 50) with higher scores indicating worse outcome (higher fatigue)
Depression using DASS-21 | Baseline, after treatment (1 week later)
  DASS-21 depression scale with cut off scores: 0-9 normal, 10-13 mild, 14-20 moderate, 21-27 severe and 28+ extremely severe
Anxiety using DASS-21 | Baseline, after treatment (1 week later)
  DASS-21 anxiety scale with cut off scores: 0-7 normal, 8-9 mild, 10-14 moderate, 15-19 severe and 20+ extremely severe
Stress using DASS-21 | Baseline, after treatment (1 week later)
  DASS-21 stress scale with cut off scores: 0-14 normal, 15-18 mild, 19-25 moderate, 26-33 severe and 34+ extremely severe
Functionality using EQ-5D-5L | Baseline, after treatment (1 week later)
  EQ-5D-5L score is from 0-100 with higher scores indicating better outcome (higher functionality)

CONTACTS AND LOCATIONS:
Locations (1):
- Cyprus University of Technology, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be available in Open Science Framework (OSF) and to anyone with reasonable request per Open Science principles.